CLINICAL TRIAL: NCT02055430
Title: Ureteral Stents Versus Percutaneous Nephrostomy for Initial Urinary Drainage in Children With Obstructive Anuria and Acute Renal Failure Due to Ureteral Calculi: a Prospective, Randomized Study
Brief Title: Ureteral Stents Versus Percutaneous Nephrostomy for Initial Urinary Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohammed said elsheemy, Associte professor of urology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61177
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Children; Obstructive Uropathy; Acute Renal Failure; Ureteric Stones
Keywords: anuria; children; nephrostomy; stents; urinary calculi
MeSH Terms: conditions — Acute Kidney Injury; Anuria; Urinary Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- percutaneous nephrostomy (Active Comparator): percutaneous nephrostomy insertion (6-8 Fr in size) for initial urinary drainage followed by definitive stone management.
  Interventions: Procedure: percutaneous nephrostomy insertion; Procedure: Definitive stone management
- Bilateral double J ureteric stents (Active Comparator): double J ureteric stent insertion (4.8-6 Fr JJ in size) for initial urinary drainage followed by definitive stone management.
  Interventions: Procedure: bilateral double J ureteric stent; Procedure: Definitive stone management

INTERVENTIONS:
Procedure: percutaneous nephrostomy insertion — The 1st arm was drained by PCN. This was performed under general anesthesia (GA) and fluoroscopic guidance.
  Other Names: PCN insertion; nephrostomy insertion
  Arms: percutaneous nephrostomy
Procedure: bilateral double J ureteric stent — The 2nd arm was drained by bilateral JJ . This was performed under general anesthesia (GA) and fluoroscopic guidance.
  Other Names: JJ
  Arms: Bilateral double J ureteric stents
Procedure: Definitive stone management — (shockwave lithotripsy, chemodissolution therapy, ureteroscopy or open surgery) for clearance of stones.
  Other Names: DSM

SUMMARY:
To compare percutaneous nephrostomy (PCN) versus double J stent (JJ) as an initial urinary drainage in children

DETAILED DESCRIPTION:
To compare percutaneous nephrostomy (PCN) versus double J stent (JJ) as an initial urinary drainage in children with obstructive calcular anuria and acute renal failure due to ureteric calculi to identify selection criteria for initial urinary drainage method to improve drainage, to decrease complications and to facilitate subsequent definitive clearance of stones as this comparison is lacking in literature

ELIGIBILITY:
Inclusion Criteria:

* children ≤12 years old presenting with Obstructive Anuria and Acute Renal Failure due to bilateral ureteric stones

Exclusion Criteria:

* Patients with grade 0-1 hydronephrosis
* fever, pyonephrosis or sepsis.
* any contraindication to both methods of drainage (urinary diversion, urethral stricture or uncontrolled coagulopathy).

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S ElSheemy, A professor, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

REFERENCES:
- [Derived] ElSheemy MS, Shouman AM, Shoukry AI, ElShenoufy A, Aboulela W, Daw K, Hussein AA, Morsi HA, Badawy H. Ureteric stents vs percutaneous nephrostomy for initial urinary drainage in children with obstructive anuria and acute renal failure due to ureteric calculi: a prospective, randomised study. BJU Int. 2015 Mar;115(3):473-9. doi: 10.1111/bju.12768. Epub 2014 Oct 20. PMID 24698195

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Percutaneous Nephrostomy | Bilateral Double J Ureteric Stents
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: the double J arm contains 90 ureterorenal units
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Nephrostomy | Bilateral Double J Ureteric Stents | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.78 (2.295) | 4.07 (2.093) | 4.42 (2.213)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 30 | 34 | 64
Region of Enrollment [Number; unit: participants]
  Egypt | 45 | 45 | 90
creatinine [Mean (Standard Deviation); unit: mg/dL] | 4.3 (1.8) | 4.8 (1.9) | 4.59 (1.901)
hydronephrosis [Number; unit: participants] — Hydronephrosis was graded according to the Society for Fetal Urology grading system for hydronephrosis
  Fernbach SK, Maizels M, Conway JJ. Ultrasound grading of hydronephrosis: introduction to the system used by the Society for Fetal Urology. PediatrRadiol 1993;23:478-80.
  participants
    grade 2 | 27 | 30 | 57
    grade 3-4 | 18 | 15 | 33
size of stone [Mean (Standard Deviation); unit: mm] | 15.011 (4.22) | 13.25 (5.37) | 14.1 (5.2)
site of stone (180 ureterorenal units) [Number; unit: ureterorenal units of participants] — each arm contains 90 ureterorenal units in 45 participants
  ureterorenal units of participants
    upper ureter | 37 | 37 | 74
    middle ureter | 16 | 15 | 31
    lower ureter | 37 | 38 | 75
radiolucency of stones [Number; unit: participants]
  patients with radiolucent stones | 27 | 28 | 55
  patients with radioopaque stones | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Period to Return to Normal Creatinine
Description: period required for normalization of serum creatinine after initial urinary drainage using percutaneous nephrostomy or ureteric stent in children with obstructive calcular anuria and Acute Renal Failure
  serum creatinine was compared to normal values in matched healthy children
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Percutaneous Nephrostomy | Bilateral Double J Ureteric Stents
Number analyzed (Participants) | 45 | 45
days | 2.22 (0.765) | 2.18 (0.777)

2. Primary Outcome: Complications of Each Drainage Method
Description: complications of initial urinary drainage using percutaneous nephrostomy or ureteric stent in children with Obstructive Anuria and Acute Renal Failure (mucosal complications, failure of insertion, slippage, fever and infection, hematuria, leakage)
  complications were calculated per 45 ureterorenal units in PCN group and 90 ureterorenal units in Double J group
Time Frame: 1 week
Reporting Status: Not Posted

3. Secondary Outcome: The Number of Subsequent Interventions Needed for Clearance of Stones .
Description: The number of subsequent interventions needed for clearance of stones after normalization of serum creatinine in relation to initial urinary drainage method using percutaneous nephrostomy or ureteric stent in children with Obstructive Anuria and Acute Renal Failure
Time Frame: 6 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Factors Affecting the Outcome of Each Group (Operative Time, Safety and Efficacy)
Description: age, site of stones, size of stones, degree of hydronephrosis
  they were calculated per 45 ureterorenal units in PCN group and 90 ureterorenal units in Double J group
Time Frame: 1 week
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Percutaneous Nephrostomy | Bilateral Double J Ureteric Stents
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 2/45 | 1/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Percutaneous Nephrostomy (N=45) | Bilateral Double J Ureteric Stents (N=45)
Fever (Renal and urinary disorders) | 2 | 1 — febrile urinary tract infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes